CLINICAL TRIAL: NCT02613221
Title: A Phase I/II Study for the Safety and Efficacy of Panitumumab in Combination With TAS-102 for Patients With RAS (KRAS, NRAS) Wild-type, Unresectable, Advanced/Recurrent Colorectal Cancer
Brief Title: A Phase I/II Study for the Safety and Efficacy of Panitumumab in Combination With TAS-102 for Patients With Colorectal Cancer
Acronym: APOLLON
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Panitumumab-1501; U1111-1176-3692 (Other: WHO); JapicCTI-153076 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2015-11-20; First posted 2015-11-24 (Estimated); Results first posted 2019-06-24 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Colorectal Cancer
Keywords: Metastatic colorectal cancer, Panitumumab, TAS-102
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Panitumumab; trifluridine tipiracil drug combination; tipiracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- panitumumab + TAS-102 combination therapy (Experimental): Panitumumab 6 mg/kg every 2 weeks, plus TAS-102 35 mg/m² given orally twice a day in 5 days followed by a 2-day rest period for 2-week cycle, and then a 14-day rest period (28 days per 1 course).
  Interventions: Drug: Panitumumab + TAS-102

INTERVENTIONS:
Drug: Panitumumab + TAS-102 — panitumumab + TAS-102 combination therapy
  Other Names: Panitumumab + Triflridine/Tipiracil (FTD/TPI)

SUMMARY:
The purpose of this study is to evaluate the combination of panitumumab and Triflridine/Tipiracil (FTD/TPI; TAS-102) in patients with RAS wild-type metastatic colorectal cancer (CRC) refractory to standard chemotherapy (oxaliplatin, fluoropyrimidines, irinotecan and angiogenesis inhibitors).

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the combination of panitumumab and TAS-102 in patients with RAS wild-type metastatic colorectal cancer (CRC) refractory to standard chemotherapy (oxaliplatin, fluoropyrimidines, irinotecan and angiogenesis inhibitors).

Patients who are judged eligible for the study based on the inclusion and exclusion criteria will be received panitumumab (6 mg/kg) every 2 weeks and TAS-102 (35 mg/m² given orally twice a day in a 28-day) in 2-week cycle of 5 days of treatment followed by a 2-day rest period, and then a 14-day rest period.

A maximum of 58 participants will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Investigator and subinvestigator judge a candidate is understand clinical trial and comply this protocol.
2. Participants who have given written consent to take part in the study after detailed explanation of the study prior to enrollment
3. Aged ≥20 to <75 years at the time of informed consent
4. Participants with unresectable adenocarcinoma originating in the large intestine (excluding carcinoma of the appendix and anal canal cancer)
5. Participants with lesion(s) that can be evaluated. It is essential to be evaluated the tumor according to the Response Evaluation Criteria in Solid Tumors (RECIST) ver. 1.1.
6. Participants who have received chemotherapies for metastatic colorectal cancer and are refractory to or failing those chemotherapies* including; fluoropyrimidines, irinotecan, oxaliplatin, and an angiogenesis inhibitors.

   *: Refractory to or failing those chemotherapies are defied as following;
   * If recurrence is observed by imaging during neoadjuvant/adjuvant therapy, or within 6 months of the completion of adjuvant therapy.
   * If imaging or clinical progression is observed during or within 3 months of the last dose of chemotherapy for advanced cancer.
   * When it is determined that the drugs (ie, fluropyrimidines, oxaliplatin, irinotecan, and angiogenesis inhibitors) are not allowed to be resume due to intolerable AE toxicities (eg, serious allergic reaction and accumulative neuropathy).
7. Participants classified as KRAS/NRAS wild-type** by KRAS/NRAS testing*.

   *: KRAS/NRAS test will be performed using the in vitro diagnostic listed in the National Health Insurance.

   **: Participants with no mutation in any of the codons shown below are considered wild type.

   KRAS: EXON2 (codon 12, 13), EXON3 (codon 59, 61), EXON4 (codon 117, 146) NRAS：EXON2 (codon 12, 13), EXON3 (codon 59, 61),EXON4 (codon 117, 146)
8. Participants are able to take medications orally.
9. Participants who satisfy the following criteria for the major organ function in tests performed within 14 days prior to enrollment

   * Neutrophil count ≥1.5×10^3/µL
   * Platelet count ≥1.0×10^4/µL
   * Hemoglobin ≥8.0 g/dL
   * Total bilirubin ≤1.5 mg/dL
   * Aspartate aminotransferase (AST) ≤ 100 IU/L ( ≤200 IU/L if liver metastases are present)
   * Alanine aminotransferase (ALT) ≤ 100 IU/L ( ≤200 IU/L if liver metastases are present)
   * Serum creatinine ≤ 1.5 mg/dL
10. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1
11. Life expectancy of ≥ 3 months (90 days) after enrollment

Exclusion Criteria:

1. Has received anti-EGFR antibodies (cetuximab or panitumumab), regorafenib, or TAS-102.
2. Has had treatment with radiotherapy and/or chemotherapy within 2 weeks (14 days) prior to study drug administration (except for limited field radiation in order to rescue of pain).
3. Known brain metastasis or strongly suspected of brain metastasis
4. Synchronous cancers or metachronous cancers with a disease-free period of ≥ 5 years (excluding colorectal cancer) excluding mucosal cancers cured or be possibly cured by regional resection (esophageal, stomach, and cervical cancer, non-melanoma skin cancer, bladder cancer, etc.).
5. Body cavity fluid that requires treatment (pleural effusion, ascites, pericardial effusion, etc.)
6. Participants who do not want to use contraception to prevent pregnancy, and women who are pregnant or breast-feeding, or test positive for pregnancy
7. Any investigational agent received within prior 4 weeks (28 days).
8. Disease requiring systemic steroids for treatment (excluding topical steroids)
9. History or obvious and extensive CT findings of interstitial pulmonary disease (interstitial pneumonia, pulmonary fibrosis, etc.)
10. Intestinal paralysis, gastrointestinal obstruction, or uncontrollable diarrhea (incapacitating symptoms despite adequate treatment.
11. Serious drug hypersensitivity (without allergy to oxaliplatin)
12. Local or systemic active infection requiring treatment, or fever indicating infection
13. NYHA class II or higher heart failure or serious heart disease
14. Active hepatitis B
15. Known HIV infection
16. Adverse event due to previous treatment that has not recovered to Grade 1 (Grade 2 for peripheral sensory neuropathy) by CTCAE (Japanese edition JCOG version 4.03) (excluding hemoglobin content)
17. Known BRAF mutation
18. Other participants judged by the investigator or subinvestigator to be ineligible for enrollment in the study (such as patients who were coerced to give consent)

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2015-12-07 (Actual); Primary Completion 2017-10-06 (Actual); Study Completion 2018-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (32):
- Japan (32):
  - Nagoya, Aichi-ken
  - Kashiwa, Chiba
  - Matsuyama, Ehime
  - Kitakyushu, Fukuoka
  - Kurume, Fukuoka
  - Hakodate, Hokkaido
  - Kushiro, Hokkaido
  - Sapporo, Hokkaido
  - Amagasaki, Hyōgo
  - Kobe, Hyōgo
  - Tsukuba, Ibaragi
  - Kasama, Ibaraki
  - Hiragi, Kagawa-ken
  - Sagamihara, Kanagawa
  - Ōsaki, Miyagi
  - Matsumoto, Nagano
  - Sasebo, Nagasaki
  - Yamatotakada, Nara
  - Takatsuki, Osaka
  - Shinden, Saitama
  - Shizuoka, Shizioka
  - Nakatogari, Shizuoka
  - Koto-ku, Tokyo
  - Minato-ku, Tokyo
  - Chiba
  - Fukui
  - Fukuoka
  - Kumamoto
  - Okayama
  - Okinawa
  - Osaka
  - Toyama

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 25 investigative sites in Japan, from 08 December 2015 to 30 March 2018.
Pre-assignment Details: Participants with a historical diagnosis of RAS wild-type, unresectable, advanced/recurrent colorectal cancer were enrolled in this study.
Groups:
- Panitumumab + TAS-102: Panitumumab 6 mg/kg every 2 weeks, plus TAS-102 35 mg/m² given orally twice a day in 5 days followed by a 2-day rest period for 2-week cycle, and then a 14-day rest period (28 days per 1 course).
Period: Overall Study
Arm/Group | Panitumumab + TAS-102
Started | 56
Safety Population: Received Study Drug | 55
Completed | 1
Not Completed | 55
Not completed — Lack of efficacy (exacerbation) | 50
Not completed — Adverse Event | 2
Not completed — Voluntary Discontinuation | 1
Not completed — Delayed Treatment | 1
Not completed — Enrolled but Not Treated | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set, The safety analysis set was defined as all participants who received at least one dose of the study drug during the study.
Arm/Group | Panitumumab + TAS-102
Number analyzed (Participants) | 55
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.5 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 29
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: Participants]
  Japan | 55
Height [Mean (Standard Deviation); unit: Centimeters (cm)] | 162.5 (9.2)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 62.66 (14.67)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] — Body Mass Index = weight (kg)/[height (m)^2]
  kilogram per square meter (kg/m^2) | 23.57 (4.39)
Duration of First-line Treatment [Median (Full Range); unit: Days] — Reported data were mean duration between the date of initiation of first-line treatment and the date of enrollment of this study.
  Days | 595.5 [72 to 2240]
Primary Tumor Location (Single/Multiple) [Count of Participants; unit: Participants] — Reported data were number of participants with primary tumor location categorized by Single or Multiple at the start of this study.
  Participants
    Single | 54
    Multiple | 1
Primary Tumor Location (Colon/Rectal) [Count of Participants; unit: Participants] — Reported data were number of participants with primary tumor location categorized by Colon or Rectal at the start of this study.
  Participants
    Colon | 34
    Rectal | 21
Primary Tumor Location (Right side/Left side) [Count of Participants; unit: Participants] — Reported data were number of participants with primary tumor location categorized by Right side or Left side at the start of this study.
  Participants
    Right side | 7
    Left side | 48
Number of metastatic organ [Count of Participants; unit: Participants]
  1 | 23
  =>2 | 32
Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) [Count of Participants; unit: Participants] — ECOG-PS is measured on 6-point scale to assess participant's performance status. 0=Fully active (best), able to carry on all pre-disease activities without restriction; 1=Restricted in physically strenuous activity, but ambulatory and able to carry out light or sedentary work; 2=Ambulatory (>50% of waking hours), capable of all selfcare, but unable to carry out any work activities; 3=Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours; 4=Completely disabled, cannot carry on any selfcare, totally confined to bed or chair; 5=Dead (worst).
  Participants
    0 | 38
    1 | 17
Resection of Primary Tumor [Count of Participants; unit: Participants] — Reported data were the number of participants who experienced resection of primary tumor. Yes; Had experienced, No; Had not experienced.
  Participants
    Yes | 43
    No | 12
Adjuvant Chemotherapy [Count of Participants; unit: Participants] — Reported data were the number of participants who experienced adjuvant chemotherapy. Yes; Had experienced, No; Had not experienced.
  Participants
    Yes | 16
    No | 39
Number of prior lines of chemotherapy [Count of Participants; unit: Participants] — Reported data were the number of participants who experienced 1, 2, or 3 prior lines of chemotherapy before the start of this study.
  Participants
    1 | 6
    2 | 37
    3 | 12
Complication [Count of Participants; unit: Participants] — Complications defined as a disease or a health condition for each participant at the start of study. Complications were classified as congenital anomalies, endocrine disorders, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, gastrointestinal (GI) disorders, renal disease and other complications. Other complications included all complications except for those mentioned above.
  Participants
    Had No Presence of Complications | 10
    Had Presence of Complications | 45

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicity (DLT) With Panitumumab Plus TAS-102 Combination Therapy
Description: DLT was evaluated according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 and was defined as any of the following events: 1. Grade 4 neutropenia for more than 7 days under maximum supportive therapy; 2. Febrile neutropenia; 3. Platelet counts decreased of Grade 3 requiring platelet transfusion or blood platelet decreased of Grade 4; 4. If Course 2 was not initiated within 14 days due to AE related to the protocol treatment; 5. Grade 3 or higher non-hematologic toxicity that was considered clinically significant, except the following cases, Grade 3 gastrointestinal symptoms that could be controlled with supportive therapy (eg, appropriate use of antiemetics, antidiarrheals), and Grade 3 or higher electrolyte abnormalities that were not deemed clinically significant.
Time Frame: Up to approximately 1 month
Population: DLT Evaluation Set; DLT Evaluation Set was defined as participants who were enrolled and received at least one dose of the study drug in order to assess recommended dose of panitumumab in combination with TAS-102 (Total number of DLT Evaluation Set was 6).
Measure: Count of Participants; unit: Participants
Arm/Group | Panitumumab + TAS-102
Number analyzed (Participants) | 6
Participants | 0

2. Primary Outcome: Progression Free Survival (PFS) Rate at 6 Months
Description: PFS rate at 6 months was defined as the crude rate of surviving participants who survived or were not determined as progressive at 6 months from the day of enrollment. Although the subjects who had no imaging data on progression at 6 months after enrollment or the subjects who had lost to follow-up were included in the denominator, these subjects were not handled as progression-free. Progression included both progression disease (PD) based on diagnostic imaging assessed according to response evaluation criteria in solid tumors (RECIST) ver 1.1 and primary disease progression that cannot be confirmed by diagnostic imaging (clinical progression). PD: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study).
Time Frame: Up to 6 months
Population: Full analysis set (FAS); FAS was defined as participants who were enrolled and received at least one dose of protocol treatment (the recommended dose confirmed in the phase I part).
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Panitumumab + TAS-102
Number analyzed (Participants) | 54
Percentage of Participants | 33.3 [22.77 to 45.32]

3. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the period from the day of enrollment until death by all causes.
Time Frame: From date of enrollment until the death, assessed up to approximately 29 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Panitumumab + TAS-102
Number analyzed (Participants) | 54
Months | 14.1 [12.18 to 19.29]

4. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the period from the day of enrollment until the day of documented progression or the day of death due to all causes whichever comes earlier. Progression included both PD based on diagnostic imaging assessed according to response evaluation criteria in solid tumors (RECIST) ver 1.1 and primary disease progression that cannot be confirmed by diagnostic imaging (clinical progression). PD: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study).
Time Frame: From date of enrollment until the date of progression or death, assessed up to approximately 29 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Panitumumab + TAS-102
Number analyzed (Participants) | 54
Months | 5.8 [4.46 to 6.50]

5. Secondary Outcome: Response Rate (RR)
Description: RR was defined as the percentage of participants who had shown complete response (CR) or partial response (PR) as the best overall response in accordance with the RECIST 1.1 criteria. The best overall response was CR, followed by PR, stable disease (SD), progressive disease (PD), and not evaluable (NE). CR: disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to <10 mm. PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters as the best overall response after randomization., SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. PD: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study).
Time Frame: From date of enrollment until the end of follow-up period, assessed up to approximately 29 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Panitumumab + TAS-102
Number analyzed (Participants) | 54
Percentage of Participants | 37.0 [24.29 to 51.26]

6. Secondary Outcome: Duration of Response (DOR)
Description: DOR means that the period from the day when either CR or PR is first confirmed until the day of documented PD or the day of death due to all causes, whichever occurs earlier.
Time Frame: From date of CR or PR until the date of PD or death, assessed up to approximately 29 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Panitumumab + TAS-102
Number analyzed (Participants) | 54
Months | 4.1 [2.29 to 6.29]

7. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR was defined as the percentage of participants who had shown CR, PR, or SD as the best overall response in accordance with the RECIST version 1.1 criteria.
Time Frame: From date of enrollment until the end of follow-up period, assessed up to approximately 29 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Panitumumab + TAS-102
Number analyzed (Participants) | 54
Percentage of Participants | 81.5 [68.57 to 90.75]

8. Secondary Outcome: Time to Treatment Failure (TTF)
Description: TTF was defined as the time from the date of enrollment to the date of the decision to discontinue the protocol treatment, the date of documented progression during the protocol treatment, or the date of death from any cause, whichever had come earlier.
Time Frame: From date of enrollment until the date of the protocol treatment discontinuation, progression or death, assessed up to approximately 29 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Panitumumab + TAS-102
Number analyzed (Participants) | 54
Months | 5.8 [4.29 to 6.21]

9. Secondary Outcome: Number of Participants Reporting One or More Treatment-Emergent Adverse Events (TEAEs)
Description: Adverse events (AEs) were any unfavorable medical events encountered in a participant treated with a drug. They were not limited to the events with clear causal relationship with treatment with the concerned drug. Treatment-emergent adverse events (TEAEs) were defined as AEs that had occurred after the initiation of protocol treatment.
Time Frame: From first dose of the study drug through 30 days after the last dose of study drug or start of subsequent antineoplastic therapy, assessed up to approximately 29 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Panitumumab + TAS-102
Number analyzed (Participants) | 55
Participants | 55

ADVERSE EVENTS:
Time Frame: From first dose of the study drug through 30 days after the last dose of study drug or start of subsequent antineoplastic therapy, assessed up to approximately 29 months
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Panitumumab + TAS-102
All-Cause Mortality (participants affected / at risk) | 6/55
Serious Adverse Events (participants affected / at risk) | 13/55
Other Adverse Events (participants affected / at risk) | 54/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Panitumumab + TAS-102 (N=55)
Anaemia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 5
Vomiting (Gastrointestinal disorders) | 1
General physical health deterioration (General disorders) | 1
Pyelonephritis (Infections and infestations) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Female genital tract fistula (Reproductive system and breast disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Device breakage (Product Issues) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Panitumumab + TAS-102 (N=55)
Anaemia (Blood and lymphatic system disorders) | 9
Vertigo (Ear and labyrinth disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 6
Diarrhoea (Gastrointestinal disorders) | 17
Nausea (Gastrointestinal disorders) | 23
Stomatitis (Gastrointestinal disorders) | 39
Vomiting (Gastrointestinal disorders) | 8
Fatigue (General disorders) | 27
Malaise (General disorders) | 10
Pyrexia (General disorders) | 9
Blood bilirubin increased (Investigations) | 4
Neutrophil count decreased (Investigations) | 36
Platelet count decreased (Investigations) | 13
White blood cell count decreased (Investigations) | 7
Hypomagnesaemia (Metabolism and nutrition disorders) | 12
Decreased appetite (Metabolism and nutrition disorders) | 30
Proteinuria (Renal and urinary disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 4
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 34
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 14
Dry skin (Skin and subcutaneous tissue disorders) | 27
Pruritus (Skin and subcutaneous tissue disorders) | 9
Rash (Skin and subcutaneous tissue disorders) | 11
Constipation (Gastrointestinal disorders) | 4
Paronychia (Infections and infestations) | 23
Back pain (Musculoskeletal and connective tissue disorders) | 5
Dysgeusia (Nervous system disorders) | 12
Peripheral sensory neuropathy (Nervous system disorders) | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-07-10): https://cdn.clinicaltrials.gov/large-docs/21/NCT02613221/SAP_000.pdf
  • Study Protocol (2017-09-29): https://cdn.clinicaltrials.gov/large-docs/21/NCT02613221/Prot_001.pdf